CLINICAL TRIAL: NCT06721273
Title: The Effect of Iodine Supplementation on Fertility Parameters in Women Experiencing Infertility
Brief Title: Iodine Supplementation and Fertility Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1402-4-418-69386
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Infertility (IVF Patients)
MeSH Terms: conditions — Infertility | interventions — Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine supplement (Experimental): In intervention group women will take 150 µg daily (one tablet per day, Tavan Institute, Tehran, Iran) that will be 2 months before starting the new in vitro fertilization (IVF) cycle.
  Interventions: Dietary Supplement: Iodine
- Placebo (Placebo Comparator): Women will take a placebo tablet daily (containing white wheat flour, which is similar to iodine table in terms of size, shape, and color, Tavan Institute, Tehran, Iran) 2 months before starting the new IVF cycle.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Iodine — In intervention group women will take 150 µg daily (one tablet per day, Tavan Institute, Tehran, Iran) that will be 2 months before starting the new in vitro fertilization (IVF) cycle.
  Arms: Iodine supplement
Dietary Supplement: Placebo — Women will take a placebo tablet daily (containing white wheat flour, which is similar to iodine table in terms of size, shape, and color, Tavan Institute, Tehran, Iran) 2 months before starting the new IVF cycle.
  Arms: Placebo

SUMMARY:
Iodine has been identified as a potential factor influencing female fertility during the childbearing years. The American Thyroid Association recommends that women attempting to conceive take a supplement containing 150 µg of iodine. However, no clinical trials have specifically examined the necessity of iodine supplementation in women experiencing infertility. Furthermore, no information is available on the optimal dose and duration of iodine supplementation to increase the chances of successful treatment in this group of women. Therefore, this study aims to investigate the effects of iodine supplementation on fertility parameters in infertile women.

DETAILED DESCRIPTION:
This double-blind randomized clinical trial will be conducted in infertility clinic on women with diminished ovarian reserve and undergoing in vitro fertilization (IVF) cycle treatment. According to the Bologna criteria, decreased ovarian reserve is defined as having 3 to 5 antral follicles and an anti-Müllerian hormone concentration ranging from 0.1 to 1.5 ng/ml. All women diagnosed with diminished ovarian reserve who meet the inclusion and exclusion criteria outlined in the general information section of the clinical trial and have provided written consent to participate will be examined. Following enrollment and baseline measurements, women will be randomly assigned to treatment groups-placebo and iodine supplement (150 µg/day of iodine)-in a 1:1 allocation ratio, using a random number table. In the intervention group, women will take 150 µg of iodine daily (one tablet per day, Tavan Institute, Tehran, Iran) for two months prior to starting the new IVF cycle. In the control group, participants will take a placebo tablet daily (containing white wheat flour, designed to match the size, shape, and color of the iodine tablet, Tavan Institute, Tehran, Iran) for the same duration before beginning the new IVF cycle. Women of two groups will be followed until the end of IVF cycle. Women in both groups will be monitored until the completion of the IVF cycle. Throughout the study, the following parameters will be assessed based on the timeline of the IVF cycle: the number of retrieved oocytes, the number of mature (MII) oocytes, the number of embryos, embryo quality, biochemical pregnancy, and clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women with diminished ovarian reserve
* Willingness to participate
* Age range: 18 to 45 years
* Women with a menstrual cycle of 21 to 42 days
* Women who have not used any contraceptive methods in the past 12 months
* Women who have not had in sexual intercourse for more than 2 months

Exclusion Criteria:

* Unwillingness to participate
* Women with polycystic ovary syndrome or endometriosis
* Diagnosis of any thyroid disease
* Use of any medication that affects the thyroid function
* Use of dietary supplements containing iodine (excluding those considered in the present study)
* Use of iodine-containing disinfectants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 230 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved oocytes | 2 weeks after the start of ovarian stimulation (approximately 2 months after intervention)
  Total count of mature eggs (oocytes) collected from a woman's ovaries during an IVF cycle through the egg retrieval procedure by embryologists
Number of mature (MII) oocytes | 2 weeks after the start of ovarian stimulation (approximately 2 months after intervention)
  Total count of oocytes that have reached the metaphase II stage of meiosis. This measurement is done by embryologists

SECONDARY OUTCOMES:
Number of embryos | 16-18 hours after insemination
  Number of fertilized eggs (oocytes) that develop into embryos after the fertilization process with sperm
Quality of embryos | 3 days after fertilization
  Quality of embryos is graded by embryologists using 3-point score scale
Biochemical pregnancy | 12 days after embryo transfer
  Biochemical pregnancy is confirmed by βHCG test
Clinical pregnancy | 3 weeks after embryo transfer
  Presence of one or more gestational sacs during transvaginal scans

IPD SHARING:
Plan to Share IPD: Undecided